CLINICAL TRIAL: NCT03478098
Title: The Importance of Glycaemic Index and Exercise on Postprandial Glucose Excursions and Gut Hormone Secretion Following Roux-en-Y Gastric Bypass
Brief Title: Meal Glycaemic Index and Exercise After Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirstine Nyvold Bojsen-Moeller (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Kirstine Nyvold Bojsen-Moeller, Kirstine Nyvold Bojsen-Moeller, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ExRYGB
Record Dates: First submitted 2018-02-06; First posted 2018-03-27 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Roux-en-Y Gastric Bypass; Obesity
Keywords: Gut hormones; Glucose excursions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 Roux-en-Y Gastric Bypass patients (Experimental): 4 study days in randomized order are conducted with interventions: Low GI mealtest, High GI mealtest, Low GI mealtest and subsequent exercise, High GI mealtest and subsequent exercise
  Interventions: Other: Low GI mealtest; Other: Low GI mealtest and subsequent exercise; Other: High GI mealtest; Other: High GI mealtest and subsequent exercise
- 10 control subjects (Experimental): 4 study days in randomized order are conducted with interventions: Low GI mealtest, High GI mealtest, Low GI mealtest and subsequent exercise, High GI mealtest and subsequent exercise
  Interventions: Other: Low GI mealtest; Other: Low GI mealtest and subsequent exercise; Other: High GI mealtest; Other: High GI mealtest and subsequent exercise

INTERVENTIONS:
Other: Low GI mealtest — Meal with low glycaemic index (GI) is consumed over 20 min
Other: Low GI mealtest and subsequent exercise — Meal with low glycaemic index (GI) is consumed over 20 min and the subject postprandially exercises for 30 min
Other: High GI mealtest — Meal with high glycaemic index (GI) is consumed over 20 min
Other: High GI mealtest and subsequent exercise — Meal with high glycaemic index (GI) is consumed over 20 min and the subject postprandially exercises for 30 min

SUMMARY:
The study will evaluate postprandial glucose excursions and gut hormone secretion after ingestion of meals with different glycaemic index (GI) values (high vs low) followed by an acute bout of exercise or rest in gastric bypass operated subjects and matched control subjects.

ELIGIBILITY:
RYGB patients:

Inclusion Criteria:

* Undergone Roux-en-Y gastric bypass (RYGB) without complications at least 12 months prior to inclusion.
* Achieved > 50% Excess BMI Loss
* Weight stability (no fluctuations over ± 5 kg the last 3 months)
* HBA1c < 48 mmol/mol before and after surgery without the use of anti-diabetic medication
* The participant must be able to ingest the meals

Exclusion Criteria:

* Low hemoglobin levels (< 6.5 mM)
* Pregnancy (determined by human chorionic gonadotropin (hCG) test) or breastfeeding
* Dysregulated thyroid gland affection
* The use of medication which affects heart frequency (i.e. Beta-blockers)
* Complications following RYGB consisting of dysphagia or other problems associated with ingestion of normal foods (i.e. vomit, diarrhea or strong abdominal pain).

Control group:

Inclusion Criteria:

* Matched with the RYGB patients on gender, age (± 5 years), menopausal state (pre- versus post-menopausal) and BMI (± 3 points).
* Weight stable ( ± 5 kg during 3 months)
* HBA1c < 48 mmol/mol

Exclusion Criteria:

* Prior bariatric surgery or prior surgery in the upper gastrointestinal tract.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Impact of acute bout of exercise on nadir plasma glucose within groups for each intervention | The lowest plasma glucose concentration at 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210 OR 240 min after ingestion of meal
  Comparison of nadir plasma glucose in response to an acute bout of exercise internally in groups a) RYGB and b) control group
Impact of glycaemic index on nadir plasma glucose within groups for each intervention | The lowest plasma glucose concentration at 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210 OR 240 min after ingestion of meal
  Comparison of nadir plasma glucose in response to meals with high vs low glycaemic index internally in groups a) RYGB and b) control group

SECONDARY OUTCOMES:
Impact of acute bout of exercise on AUC glucose within groups | AUC time-concentration-curve for plasma glucose from 0, 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210, 240 min after ingestion of meal
  Comparison of plasma glucose excursions in response to an acute bout of exercise internally in groups a) RYGB and b) control group determined by differences in area under curve (AUC)
Impact of acute bout of exercise on delta-fasting-peak glucose within groups | Difference between fasting plasma glucose and highest plasma glucose at 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210, 240 min after ingestion of meal
  Comparison of plasma glucose excursions in response to an acute bout of exercise internally in groups a) RYGB and b) control group determined by delta-fasting-to-peak concentrations of glucose
Impact of glycaemic index on AUC glucose within groups | AUC time-concentration-curve for plasma glucose from 0, 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210, 240 min after ingestion of meal
  Comparison of plasma glucose excursions in response to meals with high vs low glycaemic index internally in groups a) RYGB and b) control group determined by differences in area-under-the-curve of glucose
Impact of glycaemic index on delta-fasting-peak glucose within groups | Difference between fasting plasma glucose and highest plasma glucose at 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210, 240 min after ingestion of meal
  Comparison of plasma glucose excursions in response to meals with high vs low glycaemic index internally in groups a) RYGB and b) control group determined by differences in delta-fasting-peak glucose
Impact of postprandial exercise and meal glycaemic index on glucagon-like peptide-1 (GLP-1) secretion within the groups determined by differences in AUC | AUC for time concentration curve of GLP-1 at 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  AUC GLP-1 will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on glucagon-like peptide-1 (GLP-1) secretion within the groups determined by differences in peak concentration | Highest GLP-1 at 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Peak GLP-1 will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on ghrelin secretion within the groups determined by differences in suppression from basal values | Decremental AUC for the time concentration curve of ghrelin at 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  decremental AUC of ghrelin will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on peptide YY (PYY) secretion within the groups determined by differences in AUC | AUC for time concentration curve of PYY at 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  AUC PYY will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on peptide YY secretion within the groups determined by differences in peak concentration | Highest PYY concentration at 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Peak PYY will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on glucose-dependent insulinotropic peptide (GIP) secretion within the groups determined by differences in AUC | AUC for time concentration curve of GIP at 0,10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  AUC GIP will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on glucose-dependent insulinotropic peptide (GIP) secretion within the groups determined by differences in peak concentration | Highest concentration of GIP at 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Peak GIP will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on glucagon secretion within the groups determined by differences in AUC | AUC for time concentration curve of glucagon at 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  AUC glucagon will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on blood lactate levels within the groups determined by differences in AUC | AUC of the time-concentration curve of lactate at 0, 10, 20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 150, 180, 240 min after ingestion of meal
  AUC lactate will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on blood lactate levels within the groups determined by differences in peak concentration | Highest lactate at 10, 20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 150, 180, 240 min after ingestion of meal
  Peak lactate will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on insulin secretion within the groups determined by differences in AUC | AUC of time-concentration curve of insulin 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  AUC insulin will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycemic index on insulin secretion within the groups determined by differences in peak concentration | Highest insulin at 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Peak insulin will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise within the RYGB and control group
Impact of postprandial exercise and meal glycaemic index on ad libitum food intake within the groups determined by differences in ingested amount of ad libitum meal in grams | at 240 min following ingestion of test meal
  Grams of ad libitum food intake. Food will be served at 240 minutes after fixed breakfast meal

OTHER OUTCOMES:
Between group differences in delta-fasting-to-peak glucose for each intervention | difference between fasting glucose and highest glucose concentration at 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210, 240 min after ingestion of meal
  Impact of exercise on glucose excursions between RYGB vs Control, impact of meal glycaemic index on glucose excursions between RYGB vs Control determined by differences in delta-fasting-to-peak glucose
Between group differences in delta-peak-nadir glucose for each intervention | Difference from highest plasma glucose to subsequent lowest plasma glucose at 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210, 240 min after ingestion of meal
  Impact of exercise on glucose excursions between RYGB vs Control, impact of meal glycemic index on glucose excursions between RYGB vs Control determined by differences in delta-peak-nadir glucose
Between group differences in nadir plasma glucose for each intervention | Lowest glucose at 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210, 240 min after ingestion of meal
  Impact of exercise on glucose excursions between RYGB vs Control, impact of meal glycemic index on glucose excursions between RYGB vs Control determined by differences in nadir glucose
Between group differences in delta-nadir-end glucose for each intervention | Difference from lowest glucose to end study glucose 5, 10, 15 ,20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 135, 150, 180, 210, 240 min after ingestion of meal
  Impact of exercise on glucose excursions between RYGB vs Control, impact of meal glycemic index on glucose excursions between RYGB vs Control determined by differences in delta-nadir-end glucose
Between group differences in Glucagon like peptide-1 (GLP-1) secretion for each intervention determined by differences in AUC | AUC for time concentration curve of GLP-1 at 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on GLP-1 secretion between RYGB vs Control, impact of meal glycemic index on GLP-1 secretion between RYGB vs Control determined by differences in AUC.
Between group differences in Glucagon like peptide-1 (GLP-1) secretion for each intervention determined by differences in peak concentration | Highest GLP-1 at 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on GLP-1 secretion between RYGB vs Control, impact of meal glycemic index on GLP-1 secretion between RYGB vs Control determined by differences in peak concentration.
Between group differences in ghrelin secretion for each intervention determined by differences in suppression from basal values | Decremental AUC for the time concentration curve of ghrelin at 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on ghrelin secretion between RYGB vs Control, impact of meal glycemic index on ghrelin secretion between RYGB vs Control determined by differences in decremental AUC.
Between group differences in peptide YY secretion for each intervention determined by differences in AUC | AUC for time concentration curve of PYY at 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on peptide YY secretion between RYGB vs Control, impact of meal glycemic index on peptide YY secretion between RYGB vs Control determined by differences in AUC.
Between group differences in peptide YY secretion for each intervention determined by differences in peak concentration | Highest PYY concentration at 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on peptide YY secretion between RYGB vs Control, impact of meal glycemic index on peptide YY secretion between RYGB vs Control determined by differences in peak concentration
Between group differences in Glucose-dependent insulinotropic peptide (GIP) secretion for each intervention determined by differences in AUC | AUC for time concentration curve of GIP at 0,10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on GIP secretion between RYGB vs Control, impact of meal glycemic index on GIP secretion between RYGB vs Control determined by differences in AUC
Between group differences in Glucose-dependent insulinotropic peptide (GIP) secretion for each intervention determined by differences in peak concentration | Highest concentration of GIP at 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on GIP secretion between RYGB vs Control, impact of meal glycemic index on GIP secretion between RYGB vs Control determined by differences in peak concentration
Between group differences in glucagon secretion for each intervention determined by differences in AUC | AUC for time concentration curve of glucagon at 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on glucagon secretion between RYGB vs Control, impact of meal glycemic index on glucagon secretion between RYGB vs Control determined by differences in AUC
Between group differences in insulin secretion for each intervention determined by differences in AUC | AUC of time-concentration curve of insulin 0, 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on insulin secretion between RYGB vs Control, impact of meal glycemic index on insulin secretion between RYGB vs Control determined by differences in AUC
Between group differences in insulin secretion for each intervention determined by differences in peak concentration | Highest insulin at 10, 20, 30, 35, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on insulin secretion between RYGB vs Control, impact of meal glycemic index on insulin secretion between RYGB vs Control determined by differences in peak concentration
Between group differences in blood lactate levels for each intervention determined by differences in AUC | AUC of the time-concentration curve of lactate at 0, 10, 20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on blood lactate levels between RYGB vs Control, impact of meal glycemic index on blood lactate levels between RYGB vs Control determined by differences in AUC
Between group differences in blood lactate levels for each intervention determined by differences in peak concentration | Highest lactate at 10, 20, 30, 45, 60, 70, 80, 90, 100, 110, 120, 150, 180, 240 min after ingestion of meal
  Impact of exercise on blood lactate levels between RYGB vs Control, impact of meal glycemic index on blood lactate levels between RYGB vs Control determined by differences in peak concentration
Between group differences in ad libitum food intake for each intervention determined by differences in ingested amount of ad libitum meal in grams | at 240 min following ingestion of test meal
  Impact of exercise on ad libitum food intake between RYGB vs Control, impact of meal glycemic index on ad libitum food intake between RYGB vs Control determined by differences in ingested amount of ad libitum meal in grams. Food will be served at 240 minutes after fixed breakfast meal
Between group differences in blood levels of paracetamol ingested with fixed breakfast meal for each intervention determined by differences in time-to-peak | Time to highest paracetamol at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Time-to-peak paracetamol will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise between the RYGB vs control groups.
Between group differences in blood levels of paracetamol ingested with fixed breakfast meal for each intervention determined by differences peak concentration | Highest paracetamol at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240 min after ingestion of meal
  Peak paracetamol will be compared for meals with high vs low glycaemic index and with and without acute bout of exercise between the RYGB vs control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine N Bojsen-Moller, MD, PhD, Principal Investigator — Department of Endocrinology, Hvidovre Hospital
Locations (1):
- Department of Endocrinology, Hvidovre Hospital, Hvidovre, Denmark